CLINICAL TRIAL: NCT06802432
Title: Use of Corticosteroids on Prophylaxis of New-onset Arterial Fibrillation After Cardiac Surgery
Brief Title: Corticosteroids Prevent the Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman mohamed hesham elshaer, lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MS 716/2021
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Arrythmia; Anesthesia; Cardiac Surgery; Corticosteroids
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone (MP) group (Active Comparator): 42 patients, given 1 g of methylprednisolone post cardiopulmonary bypass immediately postoperative
  Interventions: Drug: 1 g of methylprednisolone (divided into 250 mg every 6h started once the patient arrived the pos-toparative ICU)
- Control group (No Intervention): 42 patients, underwent a standard cardiopulmonary bypass without any additional medications

INTERVENTIONS:
Drug: 1 g of methylprednisolone (divided into 250 mg every 6h started once the patient arrived the pos-toparative ICU) — 1 g of methylprednisolone (divided into 250 mg every 6h started once the patient arrived the pos-toparative ICU)
  Arms: Methylprednisolone (MP) group

SUMMARY:
Cardiopulmonary bypass and cardiac surgery are associated with a significant systemic inflammatory response that has been suggested playing a causative role in the development of postoperative atrial fibrillation (POAF). The goal of this study is to determine the efficacy of corticosteroids prophylaxis in preventing POAF, or length of intensive care unit (ICU) or hospital stay.

DETAILED DESCRIPTION:
Most cardiac operations are performed under cardiopulmonary bypass, however, it is well known that cardiopulmonary bypass often causes systemic inflammatory response characterized by leukocyte and high levels of C-reactive protein (CRP) complexes, as well high levels of inflammatory mediators that may contribute to postoperative complications including atrial fibrillation (AF), prolonged duration of intensive care unit (ICU) and hospital stay.

Postoperative atrial fibrillation has (POAF) been reported in 20% to 50% of patients following coronary artery bypass grafting (CABG) and is even higher after combined CABG and valve surgery.

It may increase stroke rates, trigger hemodynamic instability with heart failure and increase risk of thromboembolic complications.

The relationship between inflammation and atrial fibrillation after cardiac surgery is further strengthened by studies that showed that corticosteroid (CS) prophylaxis can reduce the occurrence of atrial fibrillation after cardiac surgery.

Corticosteroids (CS) can reduce the risk of atrial fibrillation after cardiac surgery in adults and reduce length of intensive care unit (ICU) and hospital stay.

It is a low-cost drug that can effectively inhibit inflammation, limit systemic capillary leakage syndrome and reduce organ damage, thus providing a theoretical basis for its clinical application.

However, the potential risks of CS remain controversial and inconclusive in terms of several side effects of CS such as hyperglycemia, gastrointestinal disturbances, and postoperative infections.

ELIGIBILITY:
Inclusion Criteria:

* Elective first time CABG or combined with valvular surgery.
* Use of b-adrenergic blockade.
* Normal sinus rhythm.

Exclusion Criteria:

* History of heart block
* History of previous episodes of AF or flutter
* History of peptic ulcer disease
* Permanent pacemaker
* Any documented or suspected supraventricular or ventricular arrhythmias
* Renal insufficiency (serum creatinine >20 mg/dL)
* Uncontrolled diabetes mellitus
* Systemic bacterial or mycotic infection
* Urgent or emergency surgery
* Patient underwent cardiac surgery without using cardiopulmonary bypass

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
overall occurrence of postoperative AF | during the first 72 hours after cardiac surgery

SECONDARY OUTCOMES:
length of the hospital stay | From the day of the surgery until the date of discharge from the hospital, up to 30 days.
  From the day of the surgery until the date of discharge from the hospital, which varies depending on the patient's clinical condition.
length of the ICU stay | from the day of the surgery ( postoperative ICU admission) until the time of transfer from the ICU to the surgical ward , up to 25 days.
  From the day of the surgery ( postoperative ICU admission) until the time of transfer from the ICU to the surgical ward , which varies depending on the patient's clinical condition.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elshaer, lecturer, Principal Investigator — faculty of medicine, ain shams university
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No